CLINICAL TRIAL: NCT05331794
Title: Design and Development of a New Line of Outdoor Fitness Equipment: "BIOFIT-Park" A Study on Ergonomics, Safety and Efficiency
Brief Title: Effects of Training on Outdoor Fitness Equipment for Health Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Noelia González-Gálvez, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CE111908; RTC-2017-6145-1 (Other Grant/Funding Number: Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2021-11-12; First posted 2022-04-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Healthy
Keywords: Outdoor fitness equipment; Outdoor gym; Physical fitness
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: "BIOFIT-Park" outdoor fitness equipment (Experimental): Refers to an arm that trains on the "BIOFIT-Park" line of outdoor fitness equipment that is currently under development and testing.
  Interventions: Behavioral: Training on BIOFIT-Park
- Experimental: Gym park equipment (Experimental): Refers to an arm that trains on gym park equipment
  Interventions: Behavioral: Training on gym park equipament

INTERVENTIONS:
Behavioral: Training on BIOFIT-Park — Participant will perform one strength training session on the new line of outdoor fitness equipment "BIOFIT-Park". 6 machines will be used. The training will consist of 3 sets of 15-20 repetitions, working at 60-65% RM. The execution speed will be 1x1, the rest between machines will be 20 seconds and macropauses of 90 seconds between series.
  Arms: Experimental: "BIOFIT-Park" outdoor fitness equipment
Behavioral: Training on gym park equipament — Participant will perform one strength training session on a gym park equipment. 6 machines will be used. The training will consist of 3 sets of 15-20 repetitions, working at 60-65% RM. The execution speed will be 1x1, the rest between machines will be 20 seconds and macropauses of 90 seconds between series.
  Arms: Experimental: Gym park equipment

SUMMARY:
Aging causes various changes in the body. This, together with a sedentary lifestyle, can lead to health problems such as loss of muscle mass and strength, bone mineral density and cardiovascular capacity. Therefore, it is essential to remain physically active in adulthood.

Outdoor fitness equipment offer a free and easy-to-use option for physical activity and health improvement. However, there are few studies that quantitatively evaluate the physical fitness and health improvement associated with the use of these parks.

Hence, the main objective is: 1) To evaluate the effects of training on outdoor fitness equipment on different body composition and health-related fitness parameters.

DETAILED DESCRIPTION:
Physiological, psychological and functional deterioration is associated with the aging process. It has been demonstrated that the practice of physical activity can prevent, slow or reduce this deterioration. Bio-healthy parks are an alternative for practicing physical activity outdoors and free of charge. However, there is no research that analyzes the effect of a planned training program in these parks.

Therefore, the objectives of this project are 1) To evaluate the effects of training on outdoor fitness equipment on different body composition and health-related fitness parameters.

The present project will be developed through a randomized controlled trial, with

1 experimental and 1 control group, with pre-test and post-test, with intra-group and inter-group analysis for each of the dependent variables of the study. The inclusion criteria are: (a) not having participated in a structured exercise program for at least 1 year, (b) being older than 50 years of age, and (c) being physically independent. The exclusion criteria are: (a) having musculoskeletal injuries or limitations that could affect the health and physical performance of the person; (b) being under medical prescription for taking medications that could influence physical performance; (c) not regularly attending the proposed sessions. Body composition and bone mineral density will be assessed by dual energy X-ray absorptiometry (DEXA).

Blood pressure by means of an automatic device (Colin BP 880, Inc., Tampa, FL). Strength by manual dynamometry (TKK 5401; Co., Ltd., Tokyo, Japan) and maximal isometric strength of knee extension and biceps flexion. Functional capacity will be assessed by means of the Chari stand test, gait speed, time up and go test and Short physical performance battery (SPPB), Sarcopenia will be assessed taking into account the reference values established for muscle quality (hand grip strength and chair stand test), muscle quantity (DEXA fat-free mass) and functional competence (gait speed, time up and go test, SPPB and 400 meter walk) established by the European Consensus (EWGSOP2). The Spinal Mouse device (Switzerland) will be used to assess the sagittal disposition of the spine (thoracic curve, lumbar curve and pelvic tilt) in standing and relaxed sitting. This technique is non-invasive. Health-related quality of life and satisfaction with life will be assessed by means of the SF36 and The Satisfaction with Life Scale (SWL) questionnaires. Mediterranean diet adherence will be assess with a Mediterranean diet adherence questionaire. Experimental group 1 will receive the exercise program on bio-healthy machinery with a frequency of 2 sessions per week of 55 minutes for 8 weeks. The machines used will be rider, low gemini, high gemini, walk, bottoms, flywheels circles, flywheels rotation, twin swing, surf, swing press and rowing.

Intensity will be controlled by subjective perception of effort and heart rate (Polar 420). There will be a warm-up 8-10 minutes, a main part 40-45 minutes and a return to calm 5-10 minutes. The intervention programs will be developed by a graduate in Physical Activity and Sport Sciences. The load will be progressed every 2 weeks. The control group will not perform any intervention program following their usual activity.

ELIGIBILITY:
Inclusion Criteria:

* Not present any surgery, pathology or condition that prevents the practice of physical activity or may interfere with the results of the tests.
* Do not present any acute infection in the last 2 weeks.
* Do not having carried out physical exercise similar to that performed during intervention.

Exclusion Criteria:

* Have answered "yes" to any of the items of the Physical Activity Readiness Questionnaire (PAR-Q).
* Have a medical contraindication to exercise.
* Failure to complete or attend training or measurements sessions during the intervention.
* Practice regular physical exercise outside the intervention or change habits that may influence the tests.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Rest Metabolic Rate | Pre-test
  Evaluation of resting metabolic rate through an indirect calorimetry test.
Heart Rate Variability | Pre-test and post-test
  Evaluation of changes in heart rate variability index measured via a heart rate monitor band.
Blood Pressure | Pre-test and post-test
  Non-invasive evaluation of systolic and diastolic peripheral blood pressure changes.
Counter Movement Jump Test | Pre-test and post-test
  Evaluation of explosive force in lower limb through vertical jump height in centimetres.
Knee Extension Rate of Foce Development Strength Test | Pre-test and post-test
  Evaluation of force production capacity per unit time through a dynamometer on a seated leg extension machine.
Knee Extension Strength Test | Pre-test and post-test
  Evaluation of the maximum voluntary contraction (MVC) of the quadriceps through a dynamometer on a seated leg extension machine.
Arm Curl Strength Test | Pre-test and post-test
  Evaluation of the maximum voluntary contraction (MVC) of the elbow flexor muscles through a dynamometer in standing position.
Lactate Blood Test | Pre-test and post-test
  Evaluation of serum lactate level (mmol/L) through a finger pick method
Excess Post-Exercise Oxygen Consumption Test | Post-test
  Evaluation of excess post-exercise oxygen consumption (EPOC) during the minutes following exercise sessions through indirect calorimetry.
Energy expenditure | During exercise
  Evaluation of energy expenditure of participants during exercise through indirect calorimetry
Heart rate | During exercise
  Evaluation of heart rate measured via a heart rate monitor band.
Subjective perception of effort | During exercise
  Evaluation of subjective perception of effort by ONMI-RES scale. The scale goes from 1 to 10 and the subject reports on his subjective perception of effort, with 1 being the lowest value and 10 the highest value.

SECONDARY OUTCOMES:
Sociodemographic questionnaire | Pre-test
  To define individual characteristics of participants such as age, gender or ethnicity.
Global Physical Activity Questionnaire | Pre-test
  Questionnaire to evaluate the level of physical activity performed in the daily routine. The questionnaire collects information on the time in minutes and frequency per week of moderate and vigorous physical activity, walking and sedentary activities. A greater time of physical activity and walking; and less time spent in sedentary activities would be considered a better score.
Dietary Recall Questionnaire | Pre-test
  24-hour pre-intervention dietary intake recording instrument.
Height | Pre-test
  Height will be assessed following the methodology proposed by the International Society for the Advancement of Kinathropometry (ISAK). The values will be expressed in meters.
Weight and bone weight | Pre-test
  Weight and bone weight will be performance with BIA-derived body composition measurements. It will be reported as a kilograms.
Percentaje of fat, hydration and muscle mass. | Pre-test
  Average of fat, hydration and muscle mass will be performance with BIA-derived body composition measurements. It will be reported as a percentaje.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No